CLINICAL TRIAL: NCT03315650
Title: RIVA-PCI Registry - Prospective Registry of Rivaroxaban in Patients With Atrial Fibrillation
Brief Title: Rivaroxaban in Patients With Atrial Fibrillation Undergoing PCI
Acronym: RIVA-PCI
Status: Completed | Type: Observational
Sponsor: IHF GmbH - Institut für Herzinfarktforschung (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: RIVA-PCI
Record Dates: First submitted 2017-10-10; First posted 2017-10-20 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2021-07

CONDITIONS: Non-valvular Atrial Fibrillation; Acute Coronary Syndrome; Percutaneous Coronary Intervention; Antithrombotic Therapy
Keywords: Non-valvular AF; ACS; PCI; NOAC; Rivaroxaban
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study evaluates the antithrombotic therapy in patients suffering from atrial fibrillation after stent implantation in Germany. Patients prescribed with the novel oral anticoagulant Rivaroxaban will be followed up over 14 months for their adherence to the medication schedule and for complications that occurred after index PCI.

DETAILED DESCRIPTION:
Patients suffering from non-valvular atrial fibrillation and presenting with an acute coronary syndrome require special attention with regard to antithrombotic therapy. Current guidelines recommend use of oral anticoagulation for almost all of these patients, the optimal antithrombotic strategy, however, has still to be defined. As with the use of any antithrombotic drug, clinicians need to balance the risks of ischemic stroke and thromboembolism, recurrent cardiac ischemia and/or stent thrombosis, and bleeding and haemorrhagic stroke.

A recently published randomized clinical trial (PIONEER AF) compared the combination of a novel oral anticoagulant (NOAC; Rivaroxaban) plus dual anti-platelet therapy (DAPT) with standard therapy consisting of vitamine K inhibitor plus DAPT. Patients treated with Rivaroxaban showed less incidence of bleedings, whereas ischemic complications, death or stroke were equal in the groups compared.

The RIVA-PCI Registry aims at providing an overview of the current antithrombotic treatment regimen in Germany in real life. Moreover, for patients receiving Rivaroxaban as part of their medication follow-up data with regard to their adherence to antithrombotic medication as well as complications over an interval of 14 months after index procedure will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years and capable of giving written informed consent
* Known or newly diagnosed non-valvular atrial fibrillation
* PCI with stent implantation during index hospital stay
* Written informed consent for participation in observational study (incl. telephone follow-up)
* Not simultaneously participating in any randomized trial

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive, unselected recruitment of patients fulfilling the eligibility criteria.
Sampling Method: Probability Sample
Enrollment: 1632 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2021-06-24 (Actual)

PRIMARY OUTCOMES:
Antithrombotic combination therapies (treatment patterns) in patients with non-valvular AF undergoing PCI | 18 months
  Real-life data on the prescription of antithrombotic medication for patients with atrial fibrillation after PCI

SECONDARY OUTCOMES:
Evaluation of antithrombotic medication during long-term follow-up | 14 months
  Patients receiving Rivaroxaban after index PCI are asked for their further antithrombotic medication in two telephone interviews (3 months and 14 months after index PCI)
Adverse Events during baseline and follow-up | 32 months
  Documentation of Adverse Events during baseline hospital stay (by treating physician) and during long-term follow-up (patient-reported)
Treatment adherence of patients | 14 months
  Patient-reported information on their adherence to the antithrombotic treatment strategy

CONTACTS AND LOCATIONS:
Overall Officials: Uwe Zeymer, Prof. Dr., Principal Investigator — Institut für Herzinfarktforschung (Institute for Cardiac Research)
Locations (13):
- Germany (13):
  - Kerckhoff-Klinik, Bad Nauheim
  - Segeberger Kliniken, Bad Segeberg
  - Gesundheitszentrum Bitterfeld-Wolfen, Bitterfeld-Wolfen
  - Klinikum Links der Weser, Bremen
  - Krankenhaus Buchholz, Buchholz
  - Klinikum Coburg, Coburg
  - SLK-Kliniken Heilbronn, Heilbronn
  - Städtisches Klinikum Ludwigshafen, Ludwigshafen
  - Universitätsklinikum Mannheim, Mannheim
  - Klinikum der Universität München , Campus Großhadern, Munich
  - Kreisklinikum Siegen, Siegen
  - Robert-Bosch-Krankenhaus, Stuttgart
  - Schwarzwald-Baar Klinikum, Villingen-Schwenningen

IPD SHARING:
Plan to Share IPD: No
An intermediate report summarizing the baseline data will be provided to Bayer (financial support).
  A final report summarizing baseline and follow-up data will be provided to ethical committees in Germany, to governmental authority, and to Bayer.
  Participating clinics will receive benchmarking reports (comparison of their own data with those of all other sites).
  Data will be made accessible to participating investigators for publication in journals and on conferences.

REFERENCES:
- [Derived] Zeymer U, Toelg R, Wienbergen H, Hobbach HP, Cuneo A, Bekeredjian R, Ritter O, Hailer B, Hertting K, Hennersdorf M, Scholtz W, Lanzer P, Mudra H, Schwefer M, Schwimmbeck PL, Liebetrau C, Thiele H, Claas C, Riemer T, Zahn R. Rivaroxaban in Patients With Atrial Fibrillation Who Underwent Percutaneous Coronary Intervention in Clinical Practice. Am J Cardiol. 2023 Feb 15;189:31-37. doi: 10.1016/j.amjcard.2022.11.009. Epub 2022 Dec 6. PMID 36493580